CLINICAL TRIAL: NCT03333941
Title: Continued Access Protocol: A Prospective, Multicenter, Single-Arm, Observational Study of the Safety and Clinical Performance of RES (Regenerative Epithelial Suspension) Prepared With the ReCell® Device Combined With Meshed Skin Graft in the Treatment of Acute Burn Injuries
Brief Title: Continued Access to the Recell® Device for Treatment of Acute Burn Injuries
Status: Completed | Type: Observational
Sponsor: Avita Medical (Industry)
Collaborators: Advanced Clinical Research Services, LLC (Other)
Responsible Party: Sponsor
Other Study IDs: CTP001-8
Record Dates: First submitted 2017-10-25; First posted 2017-11-07 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (1):
- RES (Regenerative Epithelial Suspension)
  Interventions: Device: ReCell® Autologous Cell Harvesting Device

INTERVENTIONS:
Device: ReCell® Autologous Cell Harvesting Device — RES (Regenerative Epithelial Suspension) derived from the use of the ReCell® device will be applied over skin grafts meshed more widely than conventional autografting.

SUMMARY:
The overall purpose of this continued access study is to allow ongoing treatment of subjects at selected investigational sites while the marketing application for the ReCell® Autologous Cell Harvesting Device is under FDA review. This is a prospective, multicenter, single-arm observational study to evaluate the safety and clinical performance of the ReCell® device when used as an adjunct to meshed autografts in patients with acute thermal burn injuries requiring skin grafting for closure.

DETAILED DESCRIPTION:
Patients 5 years or older with a total body surface area (TBSA) thermal burn injury between 5 and 50% (inclusive) who require autografting will be considered for participation in this study. RES (Regenerative Epithelial Suspension) derived from the use of the ReCell® device will be applied over skin grafts meshed more widely than conventional autografting. Healing, scar outcomes, pain and treatment-related adverse events will be evaluated at follow-up visits. Data concerning the clinical performance and safety of the ReCell device will be collected. Safety will be evaluated in terms of treatment and serious related adverse events.

Each subject will participate in up to 7 total visits (treatment visit and 6 follow-up study visits) over a period of 24 weeks. Up to 60 subjects will be enrolled and treated within this study at up to 15 institutions.

It is anticipated that enrollment will continue until PMA approval. Subject follow-up will continue until the last enrolled subject completes the 24-week visit.

ELIGIBILITY:
Inclusion Criteria:

1. The subject requires skin grafting as a result of an acute thermal burn injury (i.e., injuries caused by exposure of the skin to fire/flames, excessive heat, hot steam or water).
2. The area of total burn injury is 5-50% TBSA inclusive.
3. Area(s) requiring skin grafting at least 320 square centimeters.
4. The subject is at least 5 years of age.
5. The subject (or family, for those under 18 years of age) is willing and able to complete all follow-up evaluations required by the study protocol.
6. The subject is to abstain from any other treatment of the wound(s) for the duration of the study unless medically necessary.
7. The subject agrees to abstain from enrollment in any other interventional clinical trial for the duration of the study.
8. The subject and/or guardian are able to read and understand instructions and give informed, voluntary, written consent.

Exclusion Criteria:

1. The subject's burn injuries were caused by chemicals, electricity, and/or radioactive substances.
2. The subject is unable to follow the protocol.
3. The subject has other concurrent conditions that in the opinion of the investigator may compromise patient safety or study objectives.
4. The subject has a known hypersensitivity to trypsin or compound sodium lactate for irrigation (Hartmann's) solution.
5. Pregnant or lactating women.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Burn Unit
Sampling Method: Non-Probability Sample
Enrollment: 76 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2019-05-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Arizona Burn Center at Maricopa Integrated Health Systems, Phoenix, Arizona
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - University Medical Center, New Orleans, Louisiana
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - University of Tennessee Health Science Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | RES (Regenerative Epithelial Suspension)
Started | 76
Completed | 63
Not Completed | 13
Not completed — Lost to Follow-up | 10
Not completed — Death | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | RES (Regenerative Epithelial Suspension)
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 10
  Between 18 and 65 years | 54
  >=65 years | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (20.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 49
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 76

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Wound Healing
Description: Treatment area will be evaluated via direct visualization by the treating investigator. Complete wound closure is defined as ≥95 to100% re-epithelialization without drainage by week 8.
Time Frame: Confirmed by week 8, at two consecutive study visits at least 2 weeks apart up to 24 Weeks (e.g., at week 4 and week 8, or if a visit was missed, week 4 and week 12)
Population: Per Protocol
Measure: Number; unit: percentage of participants
Arm/Group | RES (Regenerative Epithelial Suspension)
Number analyzed (Participants) | 76
percentage of participants | 95.3

ADVERSE EVENTS:
Time Frame: 24 Weeks
Arm/Group | RES (Regenerative Epithelial Suspension)
All-Cause Mortality (participants affected / at risk) | 3/76
Serious Adverse Events (participants affected / at risk) | 16/76
Other Adverse Events (participants affected / at risk) | 39/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RES (Regenerative Epithelial Suspension) (N=76)
Non-healing Third Degree Burn R/T Caffeine Intake Capillary Constriction LL Arm Req. Add'l Grafting (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Pseudomonas Infection of Grafts (Infections and infestations) | 1 (1) — RECELL
Graft Loss Due to Immobility Over Posteriorly Located Pressure Bearing Surfaces Requiring Re-graftin (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Wound Cultures Positive for Staph Aureus Requiring Surgical Intervention (Infections and infestations) | 1 (1) — RECELL
Area of Flap Dehisced Requiring Inset of Flap Under Anesthesia (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Inpatient Surgery for Excision and Scar Release (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Graft Loss with Wound Infection (Infections and infestations) | 1 (1) — RECELL
Wound Infection Pseudomonas Aeruginosa (Infections and infestations) | 1 (1) — RECELL
Graft Failure with Wound Infection (Infections and infestations) | 1 (1) — RECELL
100% Graft Loss Right Leg (Injury, poisoning and procedural complications) | 1 (2) — RECELL
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) — NON-STUDY AREA
Colonic Perforation and Evisceration (Gastrointestinal disorders) | 1 (1) — NON-STUDY AREA
Aortic Thrombus (Cardiac disorders) | 1 (1) — NON-STUDY AREA
Deep Vein Thrombosis (Vascular disorders) | 1 (1) — NON-STUDY AREA
Stage 3 Necrotic Pressure Ulcer Right Heel (Skin and subcutaneous tissue disorders) | 1 (1) — NON-STUDY AREA
Ecoli Bacteremia (Infections and infestations) | 1 (1)
Multi-Organ Dysfunction with Acute Kidney Injury (Renal and urinary disorders) | 1
Cardiac Arrest with Return of Spontaneous Circulation (Cardiac disorders) | 1 (1)
Acute Respiratory Failure with Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute Blood Loss Anemia Secondary to Epistaxis, Gastric Bleeding Evidenced by Wheezing & Edema (Blood and lymphatic system disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Acute Blood Loss Anemia (Blood and lymphatic system disorders) | 1 (1)
Pulselessness Due to Progression of Metastatic State 4 Lung Cancer (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Ventilator Associated Pneumonia-Pseudomonas (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1)
Symptomatic Bradycardia (Cardiac disorders) | 1 (1)
Worsening Hyperglycemia (Blood and lymphatic system disorders) | 1 (1)
Ventilator Associated Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis - Wound Infection (Infections and infestations) | 1 (1)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Hospitalized for Hyperglycemia (Blood and lymphatic system disorders) | 1 (1)
Death due to Drug Overdose (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RES (Regenerative Epithelial Suspension) (N=76)
Ulnar Neuropathy of Left Upper Extremity (Vascular disorders) | 1 (1) — RECELL
Worsening of Previous Medical History of Neuropathic Pain (Vascular disorders) | 1 (1) — RECELL
Increase in Past Medical History of Acute Pain due to Burn Injury (Injury, poisoning and procedural complications) | 1 (1)
Melting Graft Wound Syndrome (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Slowly Healing Donor Sites at Distal Bilateral Lower Extremities Requring Excision (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Graft Melt Bilateral Posterior Lower Extremities (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Fall with Body Laceration of Study Treatment Area (General disorders) | 1 (1) — RECELL
Burn Injury Resulted in Exposure of Implantable Defribrillator (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Graft Failure 275 sq cm (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Graft Failure Approximately 275 Sq Cm. (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Bleeding to Surgical Site (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Graft Failure 150 sq cm (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Necrosis Left Knee (Infections and infestations) | 1 (1) — RECELL
Graft Failure 9 sq cm due to Knee Immobilizer (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Failed Graft Requiring Surgery (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Hypergranulation Tissue Left Torso (Skin and subcutaneous tissue disorders) | 1 (1) — RECELL
Bleeding (Vascular disorders) | 1 (1) — RECELL
Hypergranulation Tissue (Skin and subcutaneous tissue disorders) | 1 (1) — RECELL
Eschar Left Elbow (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Hypergranulation Tissue Knees and Calf (Skin and subcutaneous tissue disorders) | 1 (1) — RECELL
Hypergranulation Tissue Feet (Skin and subcutaneous tissue disorders) | 1 (1) — RECELL
Infection (Infections and infestations) | 1 (1) — RECELL
Graft Loss Right Breast (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Graft Loss to Right Thigh (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Graft Loss Abdomen (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Graft Loss Left Breast (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Graft Loss (R Buttock) (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Suspected Wound Infection (Right Buttock) (Infections and infestations) | 1 (1) — RECELL
Hypertrophic Scar to Back of Right Knee (Injury, poisoning and procedural complications) | 1 (1) — RECELL
Burn Site Pain (General disorders) | 7 (7) — RECELL
Itching (Skin and subcutaneous tissue disorders) | 2 (2) — RECELL
Burn Itching (Skin and subcutaneous tissue disorders) | 2 (2) — RECELL
Blood Loss Anemia (Blood and lymphatic system disorders) | 1 (1) — RECELL Treated Donor Site
Decreased Range of Motion of Bilateral Lower Extremities and Hands (Musculoskeletal and connective tissue disorders) | 1 (1) — Non-RECELL Treated Donor Site
Postoperative Pain (Injury, poisoning and procedural complications) | 1 (1) — Non-RECELL Treated Donor Site
Crusting Wounds at Right Ear, Scalp and Forehead (Skin and subcutaneous tissue disorders) | 1 (1) — Non-RECELL Treated Donor Site
Increased Delirium (Psychiatric disorders) | 1 (1) — Non-study Area
Thrombocytopenia (Increased from Prior Medical History) (Blood and lymphatic system disorders) | 1 (1) — Non-study Area
Growth in Right Eyelid (Unknown Type) (Eye disorders) | 1 (1) — Non-Study Area
Right Eye Ectropian (Eye disorders) | 1 (1) — Non-study Area
Graft Loss Right Forearm (Injury, poisoning and procedural complications) | 1 (1) — Non-study Area
Graft Loss (L Buttock) (Injury, poisoning and procedural complications) | 1 (1) — Non-study Area
Suspected Wound Infection (Left Buttock) (Infections and infestations) | 1 (1) — Non-study Area
Hypertrophic Scarring of Left Buttock (Skin and subcutaneous tissue disorders) | 1 (1) — Non-study Area
Nausea (Gastrointestinal disorders) | 3 (3) — Non-study Area
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) — Non-study Area
Indigestion (Gastrointestinal disorders) | 1 (1) — Non-study Area
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Non-study Area
Anxiety (Psychiatric disorders) | 1 (1) — Non-study Area
Insomnia (Psychiatric disorders) | 1 (1) — Non-study Area
Fluid Overload (Metabolism and nutrition disorders) | 1 (1)
Bilateral Lower Extremity Edema (General disorders) | 1 (1)
Acute Blood Loss Due to Postoperative Anemia (Injury, poisoning and procedural complications) | 1 (1)
Hypotensive Episode (Vascular disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Low Arterial Blood Pressure Postoperatively (Investigations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1)
Bacteremia Secondary to Exposed ICD Generator (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Klebsiella Pneumonia (Infections and infestations) | 1 (1)
Suspected Urinary Tract Infection (Infections and infestations) | 1 (1)
MRSA Tracheobronchitis (Infections and infestations) | 1 (1)
Fever (General disorders) | 2 (2)
Burn Site Pain (General disorders) | 4 (4)
Gas (Gastrointestinal disorders) | 1 (1)
Acid Reflux (Gastrointestinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/41/NCT03333941/Prot_SAP_002.pdf